CLINICAL TRIAL: NCT04710706
Title: Water-only Versus Water-CO2 (Hybrid) Colonoscopy Insertion Technique (WAVE): a Randomised Study
Brief Title: Water-only Versus Water-CO2 (Hybrid) Colonoscopy Insertion Technique
Acronym: WAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: v1.7 30.04.20
Record Dates: First submitted 2020-05-12; First posted 2021-01-15 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2021-08

CONDITIONS: Colon Polyp
Keywords: COLONOSCOPY; ENDOSCOPY
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water-alone colonoscopy (water exchange technique) (Active Comparator): During water-alone colonoscopy, gas insufflation (air or CO2) is not allowed during the insertion of the colonoscope to the caecum. Instead, water is used to facilitate the passage of the scope to the caecum. On withdrawal, CO2 is permitted.
  Interventions: Other: Colonoscopy insertion technique used during procedure
- Water-CO2 hybrid colonoscopy (modified water immersion technique) (Active Comparator): During water-CO2 hybrid colonoscopy, the operator has access to both water and CO2. In the left colon, predominately water is used to navigate the sigmoid. Once the splenic flexure is reached, a combination of water and CO2 is used to reach the caecum. On withdrawal, CO2 is permitted.
  Interventions: Other: Colonoscopy insertion technique used during procedure

INTERVENTIONS:
Other: Colonoscopy insertion technique used during procedure — Each arm is using a different colonoscopy insertion technique: either water-alone colonoscopy or water-CO2 colonoscopy.

SUMMARY:
The colonoscopy procedure involves insertion of a thin, flexible tube with a tiny camera inside (colonoscope) passed inside the bowel. To allow passage of the colonoscope and adequate visualisation of the lining of the bowel wall a range of techniques can be used. During colonoscopy, you can distend the colon with water, CO2 and air.

Air is no longer recommended for gas insufflation during colonoscopy as it causes pain and excess bowel distention. So the options are water and/or CO2 but it is not entirely clear which combination is the best and at what point during the colonoscopy.

In practice, a hybrid technique where both CO2 and water are used during the colonoscopy in used. Here, water is exclusively used to help navigate the sigmoid colon with air pockets suctioned and turbid water exchanged with clean water. From splenic flexure to caecum a mixture of water and CO2 is used.

The aim of this study is to assess procedure comfort and efficiency of two different colonoscopy insertion techniques: water-alone insertion of the colonoscope (gas insufflation not allowed on insertion; water exchange technique) versus water-CO2 hybrid insertion (water used predominately to splenic flexure with water/CO2 used to caecum; modified water immersion technique).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Capacity to consent

Exclusion Criteria:

* Pregnancy
* Previous bowel surgery
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2021-03-06 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Insertion time | During procedure
  Time taken to insert the colonoscope
Total procedure time | During procedure
  Time taken to insert and withdraw the colonoscope

SECONDARY OUTCOMES:
Caecal intubation rate | During procedure
  The proportion of procedures where the caecum is reached
Patient discomfort scores | Immediately after procedure
  Patients will subjectively assess discomfort scores following the procedure using a Visual Analogue Scale (VAS) which ranges from 0 to 10 where a higher score means a worse outcome.
Loop formation | During procedure
  Scopeguide appearance will be used to evaluate number of loops formed
Adenoma detection rate | 1 week after procedure with results of histology
  A measure of the number of adenomas detected during colonoscopy
Serrated polyp detection rate | 1 week after procedure with results of histology
  A measure of the number of serrated polyps detected during colonoscopy
Number of ancilliary procedures | During procedure
  The number of patient repositions and abdominal pressure episodes required during the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- St Mark's Hospital, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: No